CLINICAL TRIAL: NCT01976312
Title: A Randomized Double-masked, Phase III Study Assessing Ranibizumab Intravitreal Injections Versus Sham Control in Patients With Visual Impairment Due to Macular Edema (ME) Secondary to Central Retinal Vein Occlusion (CRVO) [Camellia]
Brief Title: Ranibizumab Intravitreal Injections Versus Sham Control in Patients With Central Retinal Vein Occlusion (CRVO)
Acronym: Camellia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002E2302
Record Dates: First submitted 2013-10-18; First posted 2013-11-05 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Central Retinal Vein Occlusion
Keywords: CRVO, macular edema, vision impairment, retinal vein occlusion, ranibizumab
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema; Vision Disorders | interventions — salicylhydroxamic acid; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab 0.5 mg (Experimental): PRN intravitreal injection
  Interventions: Drug: Ranibizumab 0.5 mg
- Sham injection (Sham Comparator): As of Month 3, ranibizumab 0.5 mg PRN intravitreal injections
  Interventions: Other: Sham injection

INTERVENTIONS:
Other: Sham injection — Sham injections referred to the imitation of an intravitreal injection using an injection syringe without needle.
  Arms: Sham injection
Drug: Ranibizumab 0.5 mg — Ranibizumab solution for injection was supplied in vials. Each vial contained ranibizumab concentration of 10mg/mL labeled as 0.5 mg/0.5 mL, corresponding to a 0.5 mg dose level. Ranibizumab was formulated as a sterile solution aseptically filled in a sterile glass vial for single use only
  Other Names: Lucentis
  Arms: Ranibizumab 0.5 mg

SUMMARY:
Provide efficacy and safety data on intravitreal injections of ranibizumab 0.5 mg in patients with visual impairment due to macular edema secondary to CRVO

ELIGIBILITY:
Inclusion Criteria for study and fellow eye:

• Patients with visual impairment secondary to central retinal vein occlusion (CRVO) with a BCVA between 24 and 73 letters in one eye and at least 35 letters in the other eye.

Exclusion Criteria:

* Pregnant or nursing women or women of child bearing potential unless using an effective contraception

  - Stroke or myocard infarction within 3 months prior to study
* History of malignancy within the past 5 years
* Uncontrolled hypertension
* Active infection or inflammation in any eye
* use of corticosteroids for at least 30 days in the last 6 months
* treatment with anti-angiogenic drugs in any eye within last 3 months
* Panretinal or focal/drid laser photocoagulation within the last 3 and 4 months respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- China (17):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- India (2):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bhubaneswar, Odisha
- Indonesia (2):
  - Novartis Investigative Site, Bandung, West Java
  - Novartis Investigative Site, Jakarta
- Philippines (2):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, San Juan City, Philippines
- Taiwan (2):
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taipei
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 253 patients were randomized to this study, 191 patients to the ranibizumab group and 62 patients to the sham group. One patient randomized to the ranibizumab group was excluded from all analyses as informed consent was obtained after first study procedures were performed. Therefore, this patient not included in randomized set.
Pre-assignment Details: This study consisted of the 3 periods (Screening period: Day -14 to Day -1; treatment period:
  Day 1 to Month 11; post-treatment period: Month 11 to Month 12). At Baseline (Visit 2, Day 1), eligible patients were randomized in a 3:1 ratio to one of the treatment arms
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Started | 190 | 62
Completed 3 Months | 186 | 60
Discontinued Study Prior to 3 Months | 4 | 2
Completed | 173 (Completed study at 12 months) | 53 (Completed study at 12 months)
Not Completed | 17 | 9
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Adverse Event | 6 | 6
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg | Sham Injection | Total
Number analyzed (Participants) | 190 | 62 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (12.64) | 54.1 (13.29) | 54.1 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 29 | 117
  Male | 102 | 33 | 135

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Visual Acuity (Letters) From Baseline to Month 1 Through Month 3
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters.
  Mean Visual Acuity was averaged over all monthly assessments from month 1 to month 3 and compared to Baseline.
Time Frame: Baseline, 3 Months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment group they had been assigned to at randomization. (MV-LOCF)=Mean value interpolation and last observation carried forward
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 62
Letters | 11.3 (10.77) | -2.7 (13.92)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Sham Injection; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Average Change of Best Corrected Visual Acuity (BCVA) From Baseline to Month 1 Through Month 12
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters. Mean Visual Acuity was averaged over all monthly assessments from month 1 to month 12 and compared to Baseline
Time Frame: Baseline, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 62
Letters | 12.4 (11.43) | 3.2 (14.62)

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA) Change From Baseline Over Time
Description: Visual acuity (VA) was assessed on both eyes during every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes the change in visual acuity at each visit compared to baseline
Time Frame: Month 1 to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 62
Letters
  Month 1 | 9.6 (10.2) | -0.9 (12.17)
  Month 2 | 11.6 (12.39) | -3.4 (16.04)
  Month 3 | 12.6 (12.01) | -3.8 (17.02)
  Month 4 | 10.7 (12.56) | 2.8 (15.26)
  Month 5 | 11.7 (12.62) | 3.9 (15.26)
  Month 6 | 12.3 (13.10) | 3.8 (17.20)
  Month 7 | 12.9 (13.36) | 5.0 (16.71)
  Month 8 | 12.4 (14.01) | 6.0 (16.01)
  Month 9 | 13.1 (15.10) | 5.6 (16.95)
  Month 10 | 13.5 (14.13) | 5.9 (16.77)
  Month 11 | 14.2 (13.15) | 6.8 (16.30)
  Month 12 | 14.5 (14.25) | 6.5 (17.10)

4. Secondary Outcome: Change From Baseline in Central-Sub-Field- Thickness (CSFT) Over Time
Description: OCT (optical coherence tomography) was used to assess CSFT (Central Sub-Field Thickness) representing the average retinal thickness of the circular area within 1 mm diameter around the foveal center.
Time Frame: Month 1 to month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 62
microns
  Month 1 | -393.7 (275.13) | -13.3 (207.55)
  Month 2 | -412.6 (297.50) | -7.9 (196.65)
  Month 3 | -433.3 (290.84) | -84.4 (274.98)
  Month 4 | -367.8 (305.26) | -364.8 (250.48)
  Month 5 | -407.0 (309.58) | -369.6 (273.92)
  Month 6 | -426.6 (294.63) | -372.3 (301.24)
  Month 7 | -421.5 (316.14) | -392.7 (288.74)
  Month 8 | -398.9 (299.67) | -405.2 (289.49)
  Month 9 | -422.1 (311.57) | -393.5 (323.50)
  Month 10 | -431.7 (300.95) | -395.2 (309.67)
  Month 11 | -438.1 (295.53) | -417.4 (288.08)
  Month 12 | -441.7 (306.53) | -416.4 (294.08)

5. Secondary Outcome: Number of Participants With a Best Corrected Visual Acuity (BCVA) Improvement of ≥5, ≥10, ≥15, and ≥30 Letters Over Time
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters.
Time Frame: Month 1 to month 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 62
Participants
  Month 1 Gain of >=5 letters | 141 | 17
  Month 1 Gain of >=10 letters | 94 | 6
  Month 1 Gain of >=15 letters | 56 | 2
  Month 1 Gain of >=30 letters | 3 | 0
  Month 2 Gain of >=5 letters | 150 | 18
  Month 2 Gain of >=10 letters | 119 | 11
  Month 2 Gain of >=15 letters | 74 | 3
  Month 2 Gain of >=30 letters | 9 | 0
  Month 3 Gain of >=5 letters | 153 | 19
  Month 3 Gain of >=10 letters | 117 | 11
  Month 3 Gain of >=15 letters | 76 | 4
  Month 3 Gain of >=30 letters | 12 | 0
  Month 4 Gain of >=5 letters | 138 | 31
  Month 4 Gain of >=10 letters | 107 | 21
  Month 4 Gain of >=15 letters | 68 | 11
  Month 4 Gain of >=30 letters | 14 | 2
  Month 5 Gain of >=5 letters | 143 | 34
  Month 5 Gain of >=10 letters | 116 | 23
  Month 5 Gain of >=15 letters | 80 | 13
  Month 5 Gain of >=30 letters | 13 | 1
  Month 6 Gain of >=5 letters | 147 | 39
  Month 6 Gain of >=10 letters | 121 | 28
  Month 6 Gain of >=15 letters | 87 | 12
  Month 6 Gain of >=30 letters | 14 | 13
  Month 7 Gain of >=5 letters | 152 | 37
  Month 7 Gain of >=10 letters | 121 | 29
  Month 7 Gain of >=15 letters | 91 | 14
  Month 7 Gain of >=30 letters | 14 | 3
  Month 8 Gain of >=5 letters | 143 | 39
  Month 8 Gain of >=10 letters | 127 | 28
  Month 8 Gain of >=15 letters | 95 | 19
  Month 8 Gain of >=30 letters | 16 | 3
  Month 9 Gain of >=5 letters | 147 | 40
  Month 9 Gain of >=10 letters | 126 | 26
  Month 9 Gain of >=15 letters | 94 | 17
  Month 9 Gain of >=30 letters | 17 | 3
  Month 10 Gain of >=5 letters | 152 | 39
  Month 10 Gain of >=10 letters | 128 | 29
  Month 10 Gain of >=15 letters | 95 | 16
  Month 10 Gain of >=30 letters | 18 | 4
  Month 11 Gain of >=5 letters | 153 | 40
  Month 11 Gain of >=10 letters | 134 | 29
  Month 11 Gain of >=15 letters | 101 | 19
  Month 11 Gain of >=30 letters | 18 | 4
  Month 12 Gain of >=5 letters | 151 | 39
  Month 12 Gain of >=10 letters | 131 | 30
  Month 12 Gain of >=15 letters | 99 | 21
  Month 12 Gain of >=30 letters | 24 | 3

6. Secondary Outcome: Number of Participants With Best Corrected Visual Acuity (BCVA)Loss of <15 Letters in the Study Eye Over Time
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes for each post-baseline month whether or not a patient lost less than 15 letters of VA as compared with baseline.
Time Frame: Month 1 to 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 62
Participants
  Month 1, Loss of < 15 letters | 185 | 57
  Month 2, Loss of < 15 letters | 182 | 53
  Month 3, Loss of < 15 letters | 182 | 51
  Month 4, Loss of < 15 letters | 179 | 55
  Month 5, Loss of < 15 letters | 182 | 56
  Month 6, Loss of < 15 letters | 180 | 53
  Month 7, Loss of < 15 letters | 181 | 55
  Month 8, Loss of < 15 letters | 177 | 55
  Month 9, Loss of < 15 letters | 177 | 56
  Month 10, Loss of < 15 letters | 180 | 56
  Month 11, Loss of < 15 letters | 183 | 56
  Month 12, Loss of < 15 letters | 182 | 55

7. Secondary Outcome: The Change in Patient Reported Outcomes in NEI-VFQ-25 Score (Composite Score and Subscales) at Month 3, 6 and 12 Compared to Baseline
Description: The VFQ-25 consists of 25 vision related questions across 11 vision related subscales, including general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision and peripheral vision, and a general health rating. Items are converted to a 0-100 scale on each subscale and for the composite score where higher scores represents better functioning.
Time Frame: Month 3,6 and 12
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment group they had been assigned to at randomization. n= is the number of patients with a value for both baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 190 | 62
Scores on a scale
  Month 3: number analyzed (Participants) | 186 | 61
  Month 3 | 4.4 (12.54) | 0.1 (13.78)
  Month 6: number analyzed (Participants) | 179 | 57
  Month 6 | 6.7 (15.02) | 2.9 (13.33)
  Month 12: number analyzed (Participants) | 173 | 53
  Month 12 | 8.2 (13.70) | 3.2 (15.34)

ADVERSE EVENTS:
Description: The Safety Set consisted of all patients who received at least one application of study treatment and had at least one post-Baseline safety assessment. Patients were analyzed according to the treatment received. The statement that a patient had no AEs also constituted a safety assessment.
Groups:
- Sham With Ranibizumab 0.5 mg: As of Month 3, ranibizumab 0.5 mg PRN intravitreal injections
- Sham Without Ranibizumab 0.5 mg: Sham without Ranibizumab 0.5mg(hereafter referred to as sham group up to Month 3 and sham without ranibizumab after Month 3
Arm/Group | Ranibizumab 0.5 mg | Sham With Ranibizumab 0.5 mg | Sham Without Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 11/190 | 5/56 | 1/5
Other Adverse Events (participants affected / at risk) | 96/190 | 32/56 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=190) | Sham With Ranibizumab 0.5 mg (N=56) | Sham Without Ranibizumab 0.5 mg (N=5)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 2 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=190) | Sham With Ranibizumab 0.5 mg (N=56) | Sham Without Ranibizumab 0.5 mg (N=5)
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Asthenopia (Eye disorders) | 2 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 17 | 3 | 0
Conjunctival hyperaemia (Eye disorders) | 3 | 1 | 0
Conjunctival oedema (Eye disorders) | 2 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 7 | 1 | 1
Eye discharge (Eye disorders) | 1 | 1 | 0
Eye irritation (Eye disorders) | 4 | 0 | 0
Eye pain (Eye disorders) | 4 | 2 | 1
Eye pruritus (Eye disorders) | 2 | 1 | 0
Eye swelling (Eye disorders) | 4 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 2 | 0 | 1
Iris neovascularisation (Eye disorders) | 0 | 2 | 1
Lacrimation increased (Eye disorders) | 2 | 0 | 0
Macular fibrosis (Eye disorders) | 2 | 0 | 0
Macular oedema (Eye disorders) | 1 | 3 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 9 | 2 | 0
Ocular hypertension (Eye disorders) | 2 | 4 | 0
Retinal haemorrhage (Eye disorders) | 1 | 5 | 0
Retinal ischaemia (Eye disorders) | 2 | 1 | 0
Retinal neovascularisation (Eye disorders) | 1 | 1 | 0
Retinal vein occlusion (Eye disorders) | 2 | 2 | 0
Vision blurred (Eye disorders) | 9 | 1 | 0
Visual acuity reduced (Eye disorders) | 9 | 3 | 1
Vitreal cells (Eye disorders) | 2 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 3 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 9 | 4 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 19 | 5 | 0
Pharyngitis (Infections and infestations) | 5 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0
Intraocular pressure increased (Investigations) | 10 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 11 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety